CLINICAL TRIAL: NCT02141243
Title: Randomized, Controlled Trial Evaluating Lingual Frenotomy in Newborns With Simultaneous Lip Tie for the Relief of Breastfeeding Pain.
Brief Title: Prospective Evaluation of Lingual Frenotomy in Newborns With Simultaneous Lip Tie for the Relief of Breastfeeding Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: FRENOTOMY
Record Dates: First submitted 2014-04-21; First posted 2014-05-19 (Estimated); Last update posted 2019-06-12 (Actual); Status verified 2018-05

CONDITIONS: Ankyloglossia; Breast Feeding; Enlarged Labial Frenum
MeSH Terms: conditions — Ankyloglossia; Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): All participants will receive both the lingual frenotomy and sham procedure. Group A infants will receive lingual frenotomy for intervention #1 and a sham procedure for intervention #2. Newborns that continue to have difficulty with breastfeeding after both interventions will undergo intervention #3, a labial frenotomy.
  Lingual frenotomy: tongue will be elevated, expose frenulum with a grooved director or 2 cotton tipped applicators, and then incise frenulum tissue with a straight scissor.
  Sham/placebo procedure: infant brought into a procedure room and kept there for as long as the average experimental procedure would take (~5 minutes).
  Maxillary labial frenotomy: 0.1 ml of 1% lidocaine will be injected into the area, upper lip lifted, frenum stretched, and a laser, (iLaseTM 940 ± 15 nm) or scissors, will be used to release its attachment to the level of the periosteum.
  Interventions: Procedure: Lingual Frenotomy; Procedure: Labial Frenotomy; Procedure: Sham Procedure
- Group B (Experimental): All participating infants will receive both the lingual frenotomy and sham procedure. Group B infants will receive the sham procedure for intervention #1 and a lingual frenotomy for intervention #2. Newborns that continue to have difficulty with breastfeeding after both interventions will undergo intervention #3, a labial frenotomy.
  Sham/placebo procedure: infant brought into a procedure room and kept there for as long as the average experimental procedure would take (~5 minutes).
  Lingual frenotomy: tongue will be elevated, expose frenulum with a grooved director or 2 cotton tipped applicators, and then incise frenulum tissue with a straight scissor.
  Maxillary labial frenotomy: 0.1 ml of 1% lidocaine will be injected into the area, upper lip lifted, frenum stretched, and an iLaseTM 940 ± 15 nm laser used to release its attachment to the level of the periosteum.
  Interventions: Procedure: Lingual Frenotomy; Procedure: Labial Frenotomy; Procedure: Sham Procedure

INTERVENTIONS:
Procedure: Lingual Frenotomy — For newborns receiving the ankyloglossia frenotomy, the tongue will be elevated and the frenulum exposed with a grooved director or 2 cotton tipped applicators. The frenulum tissue will then be incised with a straight scissor. If thick, it will be crushed with a straight clamp to provide anesthesia and decrease bleeding, and the exposed and previously clamped tongue frenulum will be incised with a straight scissor.
Procedure: Labial Frenotomy — For newborns receiving the maxillary labial frenotomy, 0.1 ml of 1% lidocaine will be injected into the area. The upper lip will be lifted and the frenum stretched. Then an iLaseTM 940 ± 15 nm laser will be used to release its attachment to the level of the periosteum.
Procedure: Sham Procedure — For newborns receiving the maxillary labial frenotomy, 0.1 ml of 1% lidocaine will be injected into the area. The upper lip will be lifted and the frenum stretched. Then an iLaseTM 940 ± 15 nm laser will be used to release its attachment to the level of the periosteum.

SUMMARY:
We are proposing to conduct a randomized, controlled trial of newborns in the maternal infant care areas at Tampa General Hospital. Participants who are determined eligible for the study (classified to have ankyloglossia via the HATLFF and either a Class III or IV maxillary labial frenum) will be randomly assigned to one of two groups: Group A or Group B. Group A will receive a sham procedure for intervention #1 and a lingual frenotomy procedure for intervention #2. Group B will receive a lingual frenotomy procedure for intervention #1 and a sham procedure for intervention #2. Newborns that continue to have difficulty with breastfeeding after both interventions will undergo intervention #3, a labial frenotomy, and breastfeeding will be monitored afterwards.

DETAILED DESCRIPTION:
The study is a randomized control studies which aims to contribute data to a previous study on the effects of ankyloglossia (tongue-tie) on breastfeeding, and to also provide new information on the effects of maxillary lip-tie on breastfeeding. Participants who are determined eligible for the study (classified to have ankyloglossia via the HATLFF and either a Class III or IV maxillary labial frenum) will be randomly assigned to one of two groups: Group A or Group B. Group A will receive a sham procedure for intervention #1 and a lingual frenotomy procedure for intervention #2. Group B will receive a lingual frenotomy procedure for intervention #1 and a sham procedure for intervention #2. Newborns that continue to have difficulty with breastfeeding after both interventions will undergo intervention #3, a labial frenotomy, and breastfeeding will be monitored afterwards. These results will be analyzed to determine when lingual frenotomies, labial frenotomies, or both are necessary to improve breastfeeding pain and LATCH scores.

The study aims to prove that the simple and low risk frenotomy procedure should be considered as treatment for both ankyloglossia and maxillary lip-tie, preventing breastfeeding complications as well as many other future problems such as with speech and self esteem. It is hypothesized that the use of frenotomies as treatment for ankyloglossia and maxillary lip-tie will improve breastfeeding success for breastfeeding couplets with newborns with both ankyloglossia and maxillary lip-tie. It is expected to see an increase in LATCH score to >7 for breastfeeding sessions and a significant decrease in scoring on the pain scale after frenotomy intervention, while it is expected to see little change in LATCH and pain scale assessment scores after sham procedures. Overall data is not expected to vary significantly between Group A and Group B. It is also hypothesized that a lingual frenotomy alone will be sufficient to improve breastfeeding success without the need to also conduct a labial frenotomy.

ELIGIBILITY:
Inclusion Criteria:

1. Newborn is full term (at least 37 weeks) and otherwise in good health.
2. Newborn exhibits having ankyloglossia (score of less than 11 with failing lactation management or an appearance score lower than 8, based on HATLFF) and a Class III or Class IV maxillary lip-tie, simultaneously.
3. Mother of newborn noted to have nipple pain or difficulty with breastfeeding (LATCH score of <7).
4. Mother of newborn has intention to exclusively breastfeed newborn.
5. Mother of newborn signs a written informed consent for treatment.

Exclusion Criteria:

1. Premature newborns.
2. Newborns older than 2 weeks.
3. Newborns with craniofacial anomalies (i.e. cleft lip or palate).
4. Newborns who are neurologically compromised.
5. Mother has condition that could affect the milk supply (i.e diabetes).
6. Mother of newborn is not English speaking and not able to read at least at a 6th grade level.

Max Age: 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2015-05; Primary Completion 2018-04 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Change in Wong-Baker FACES Pain Rating Scale | after breastfeeding before intervention #1, after breastfeeding after intervention #1, after breastfeeding after intervention #2, and during 1 week follow-up (also after intervention #3 if applicable)
  This visual pain analog scale is used to measure breastfeeding pain experienced by the mother.
Change in LATCH score | after breastfeeding before intervention #1, after breastfeeding after intervention #1, after breastfeeding after intervention #2, and during 1 week follow-up (also after intervention #3 if applicable)
  Latch, Audible swallowing, Type of nipple, Comfort, and Hold (LATCH) Breastfeeding Quality Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Pat Ricalde, MD, Principal Investigator — University of South Florida
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

REFERENCES:
- [Background] Dollberg S, Botzer E, Grunis E, Mimouni FB. Immediate nipple pain relief after frenotomy in breast-fed infants with ankyloglossia: a randomized, prospective study. J Pediatr Surg. 2006 Sep;41(9):1598-600. doi: 10.1016/j.jpedsurg.2006.05.024. PMID 16952598
- [Background] Kotlow L. Diagnosis and treatment of ankyloglossia and tied maxillary fraenum in infants using Er:YAG and 1064 diode lasers. Eur Arch Paediatr Dent. 2011 Apr;12(2):106-12. doi: 10.1007/BF03262789. PMID 21473843
- [Background] Segal LM, Stephenson R, Dawes M, Feldman P. Prevalence, diagnosis, and treatment of ankyloglossia: methodologic review. Can Fam Physician. 2007 Jun;53(6):1027-33. PMID 17872781
- [Background] Buryk M, Bloom D, Shope T. Efficacy of neonatal release of ankyloglossia: a randomized trial. Pediatrics. 2011 Aug;128(2):280-8. doi: 10.1542/peds.2011-0077. Epub 2011 Jul 18. PMID 21768318
- [Background] Edmunds J, Miles SC, Fulbrook P. Tongue-tie and breastfeeding: a review of the literature. Breastfeed Rev. 2011 Mar;19(1):19-26. PMID 21608523
- [Background] Gartner LM, Morton J, Lawrence RA, Naylor AJ, O'Hare D, Schanler RJ, Eidelman AI; American Academy of Pediatrics Section on Breastfeeding. Breastfeeding and the use of human milk. Pediatrics. 2005 Feb;115(2):496-506. doi: 10.1542/peds.2004-2491. PMID 15687461
- [Background] Masaitis NS, Kaempf JW. Developing a frenotomy policy at one medical center: a case study approach. J Hum Lact. 1996 Sep;12(3):229-32. doi: 10.1177/089033449601200321. PMID 9025430
- [Background] Wiessinger D, Miller M. Breastfeeding difficulties as a result of tight lingual and labial frena: a case report. J Hum Lact. 1995 Dec;11(4):313-6. doi: 10.1177/089033449501100419. PMID 8634108
- [Background] Kotlow LA. The influence of the maxillary frenum on the development and pattern of dental caries on anterior teeth in breastfeeding infants: prevention, diagnosis, and treatment. J Hum Lact. 2010 Aug;26(3):304-8. doi: 10.1177/0890334410362520. Epub 2010 Mar 22. PMID 20308621
- [Background] Bagga S, Bhat KM, Bhat GS, Thomas BS. Esthetic management of the upper labial frenum: a novel frenectomy technique. Quintessence Int. 2006 Nov-Dec;37(10):819-23. PMID 17078281
- [Background] Kotlow LA. Diagnosing and understanding the maxillary lip-tie (superior labial, the maxillary labial frenum) as it relates to breastfeeding. J Hum Lact. 2013 Nov;29(4):458-64. doi: 10.1177/0890334413491325. Epub 2013 Jul 2. PMID 23821655
- [Background] Amir LH, James JP, Donath SM. Reliability of the hazelbaker assessment tool for lingual frenulum function. Int Breastfeed J. 2006 Mar 9;1(1):3. doi: 10.1186/1746-4358-1-3. PMID 16722609
- [Background] Jensen D, Wallace S, Kelsay P. LATCH: a breastfeeding charting system and documentation tool. J Obstet Gynecol Neonatal Nurs. 1994 Jan;23(1):27-32. doi: 10.1111/j.1552-6909.1994.tb01847.x. PMID 8176525